CLINICAL TRIAL: NCT03182439
Title: Accuracy of Commercially Available Heart Rate Monitors in Cardiac Rehabilitation Patients: A Prospective, Randomized Study
Brief Title: Accuracy of Commercially Available Heart Rate Monitors III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 17-661
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Cardiac Rehabilitation
Keywords: WEARABLE HEART RATE MONITORS, ACCURACY

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fit Bit Blaze (Active Comparator): Fit Bit Blaze Heart Rate Monitoring Device
  Interventions: Device: Fit Bit Blaze; Device: Garmin Forerunner 235; Device: Tom Tom Spark Cardio; Device: Apple Watch
- Garmin Forerunner 235 (Active Comparator): Garmin Forerunner 235 Heart Rate Monitoring Device
  Interventions: Device: Fit Bit Blaze; Device: Garmin Forerunner 235; Device: Tom Tom Spark Cardio; Device: Apple Watch
- Tom Tom Spark Cardio (Active Comparator): Tom Tom Spark Cardio Heart Rate Monitoring Device
  Interventions: Device: Fit Bit Blaze; Device: Garmin Forerunner 235; Device: Tom Tom Spark Cardio; Device: Apple Watch
- Apple Watch (Active Comparator): Apple Watch Heart Rate Monitoring Device
  Interventions: Device: Fit Bit Blaze; Device: Garmin Forerunner 235; Device: Tom Tom Spark Cardio; Device: Apple Watch

INTERVENTIONS:
Device: Fit Bit Blaze — Fit Bit Blaze Heart Rate Monitoring Device
Device: Garmin Forerunner 235 — Garmin Forerunner 235 Heart Rate Monitoring Device
Device: Tom Tom Spark Cardio — Tom Tom Spark Cardio Heart Rate Monitoring Device
Device: Apple Watch — Apple Watch Heart Rate Monitoring Device

SUMMARY:
The objective of this study is to evaluate the accuracy of four heart rate monitors in cardiac rehabilitation patients during typical, supervised cardiac rehabilitation involving exercise on a treadmill and/or stationary bicycle.

DETAILED DESCRIPTION:
This study will assess the accuracy of four of the best-selling optical heart rate monitors when worn by cardiac rehabilitation patients.

During testing, each subject will wear:

1. Two different optical heart rate monitors (one on each wrist)
2. A Polar chest-strap based monitor
3. ECG leads

The types of wrist-worn heart rate monitors assigned to each subject will be randomly assigned.

The location (left or right wrist) will also be randomly assigned.

Heart rate will be assessed using each of the 4 monitors with the subject on the exercise machines under each of the following conditions:

1. Pre-exercise
2. Treadmill: at 3, 5 and 7 min.
3. Stationary Cycle: at 3, 5 and 7 min.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients enrolled in cardiac rehabilitation program at Cleveland Clinic Main Campus

Exclusion Criteria:

* Presence of a cardiac pacemaker
* Known chronic and persistent heart rhythm disorders
* Tattoos around the wrist or forearm area
* Use of a radial artery graft for coronary artery bypass grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Heart Rate Monitor Accuracy Compared to ECG | 16 minutes
  The primary outcome measure is the accuracy of each heart rate monitor compared to ECG. This will be expressed by the correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang R, Blackburn G, Desai M, Phelan D, Gillinov L, Houghtaling P, Gillinov M. Accuracy of Wrist-Worn Heart Rate Monitors. JAMA Cardiol. 2017 Jan 1;2(1):104-106. doi: 10.1001/jamacardio.2016.3340. No abstract available. PMID 27732703